CLINICAL TRIAL: NCT00116532
Title: Escitalopram for the Treatment of Obsessive Compulsive Disorder
Brief Title: Escitalopram for the Treatment of Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-P-000895; LXP-MD-14; 1200-211220
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Escitalopram; SSRI; Open Label
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
The purpose of this study is to assess the efficacy of Escitalopram in the treatment of obsessive compulsive disorder and to determine the optimal treatment dose.

DETAILED DESCRIPTION:
Background and Purpose: Obsessive compulsive disorder affects approximately 3% of the population. Treatment options include the selective serotonin reuptake inhibitors (SSRIs), dual serotonin and norepinephrine reuptake inhibitors, and behavioral therapy. A recent double-blind, placebo-controlled trial demonstrated that citalopram is effective in the treatment of OCD. Escitalopram is a new SSRI that may be more effective than other SSRIs for the treatment of major depression and may have fewer side effects. This study aims to assess the efficacy of escitalopram for the treatment of OCD.

Comparisons: Subject Y-BOCs pre-post treatment. We will also compare the improvement of subjects across the three different medication levels: 10 mg, 20 mg, and 30 mg.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD by DSM-IV
* Age 18-65
* Y-BOCS greater than 20
* Written informed consent
* Females of childbearing potential must have a negative serum or urinary beta-HCG test.

Exclusion Criteria:

* Pregnant women or women of childbearing potential who are not using a medically accepted means of contraception.
* Patients who, in the investigator's judgement, pose a serious suicidal or homicidal risk.
* Serious or unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease. Patients on anticoagulant therapy.
* History of seizure disorder
* Comorbid bipolar disorder, psychosis, organic mental disorder, or developmental disorder
* If there is a history of substance abuse, patients in remission at least 6 months.
* Currently being treated with behavioral therapy, specifically exposure and response prevention, for OCD.
* Other medications for medical disorders that may interfere with escitalopram
* Current major depression or prescribed an antidepressant for major depression within the past 12 months.
* Taken an SSRI medication within 2 weeks of beginning the study (4 weeks for fluoxetine).
* More than 1 adequate trial (at least 10 weeks at maximally tolerated dose) with another SSRI in the past.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-10; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Y-BOCs scores at 1st and last visit (16 weeks later)
Clinical Global impressions Scale at 2nd visit (2 weeks after 1st visit) and 6th visit (16 weeks post 1st visit)

SECONDARY OUTCOMES:
HAMD - first and last visit (Given week 0, 2, 4, 8, 12, & 16. Comparisons from week 0 and 16)
BDI - first and last visit (Given week 0, 2, 4, 8, 12, & 16. Comparisons from week 0 and 16)
BAI - first and last visit Given week 0, 2, 4, 8, 12, & 16. Comparisons from week 0 and 16)
QLESQ - first and last visit (week 0 and 16)

CONTACTS AND LOCATIONS:
Overall Officials: Darin D Dougherty, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital - OCD Clinic, Charlestown, Massachusetts, United States